CLINICAL TRIAL: NCT06007378
Title: Optimizing Postoperative Pain Control After Laparoscopic Colorectal Surgery by Supplementing Ultrasound-guided Erector Spinae Plane Block With Ketamine or Transdermal Fentanyl Patch
Brief Title: Optimizing Postoperative Pain Control After Laparoscopic Colorectal Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Ibrahim Mamdouh Esmat, Assistant Professor of Anesthesia and Intensive Care, Faculty of Medicine, Ain- shams University, Cairo, Egypt., Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: FMASU MS 416 / 2023
Record Dates: First submitted 2023-08-17; First posted 2023-08-23 (Actual); Last update posted 2025-07-28 (Actual); Status verified 2025-07

CONDITIONS: Postoperative Pain
MeSH Terms: conditions — Pain, Postoperative | interventions — Bupivacaine; Ketamine

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Bupivacaine and ketamine (Other)
  Interventions: Other: Bupivacaine and ketamine
- Bupivacaine and transdermal fentanyl patch (Other)
  Interventions: Other: Bupivacaine and transdermal fentanyl patch
- Bupivacaine (Other)
  Interventions: Other: Bupivacain

INTERVENTIONS:
Other: Bupivacaine and ketamine — Bilateral erector spinae plane block (bupivacaine and ketamine)
  Arms: Bupivacaine and ketamine
Other: Bupivacaine and transdermal fentanyl patch — Bilateral erector spinae plane block (bupivacaine) and transdermal fentanyl patch
  Arms: Bupivacaine and transdermal fentanyl patch
Other: Bupivacain — Bilateral erector spinae plane block (bupivacaine)
  Arms: Bupivacaine

SUMMARY:
Erector spinae plane block (ESPB) is a novel regional block technique that was proven to have superior outcomes in relieving postoperative pain in colorectal surgeries.Ketamine enhances the impact of local anaesthetics by reducing the duration and extent of motor block while shortening the onset of sensory and motor block.Transdermal Fentanyl Patch (TFP) was better than transdermal buprenorphine in postoperative analgesia following abdominal surgeries.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing laparoscopic colorectal surgery.
* American Society of Anesthesiologists (ASA) physical status I or II.

Exclusion Criteria:

* Known allergy to one of the study medications.
* Skin infections at the site of the needle puncture.
* Hepatic, renal or cardiac dysfunction.
* Patients diagnosed with obstructive sleep apnoea

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2023-09-05 (Actual); Primary Completion 2025-07-22 (Actual); Study Completion 2025-07-22 (Actual)

PRIMARY OUTCOMES:
The total rescue analgesia consumption (mg) | in the first 48 hours after surgery
  The total rescue analgesia consumption (mg) in the first 48 hours after surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Ain-Shams University Hospitals, Cairo, Egypt